CLINICAL TRIAL: NCT02347592
Title: Comparison of Self-locating Catheter Versus a Straight Catheter for Outflow Problems.
Brief Title: Peritoneal Dialysis Catheter Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Umeå (Other)
Responsible Party: Principal Investigator, Bernd Stegmayr, Professor, University Hospital, Umeå
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: UHUmea01
Record Dates: First submitted 2014-12-10; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- straight Tenckhoff (Active Comparator): The straight Tenckhoff catheter (sT) is the most common used catheter for peritoneal dialysis (PD).
  Interventions: Device: straight Tenckhoff
- self-locating catheter (Active Comparator): A new, more expensive, self-locating catheter (sLC) has been developed by Di Paolo.
  Interventions: Device: Self-locating Catheter

INTERVENTIONS:
Device: Self-locating Catheter — Procedure/Surgery necessary if obstruction occurs
  Arms: self-locating catheter
Device: straight Tenckhoff — Procedure/Surgery necessary if obstruction occurs
  Arms: straight Tenckhoff

SUMMARY:
The straight Tenckhoff is the most common catheter for peritoneal dialysis. A new, more expensive,self-locating catheter with a heavy tip has been developed by Di Paolo. The investigators used these catheters in parallel for several years. To clarify what catheter has least problems the investigators performed a comparative study to clarify if outflow problems differed between these catheters.

DETAILED DESCRIPTION:
The straight Tenckhoff catheter (sT) is the most common used catheter for peritoneal dialysis (PD). A new, more expensive, self-locating catheter (sLC) has been developed by Di Paolo. The investigators had used both in parallel for several years. To clarify what catheter to focus on in the future the investigators performed a comparative study to clarify if outflow problems differed between these catheters.

Study design: interventional and randomized at the same hospital Patients: Patients that were planned to start PD were informed and asked to participate in the randomized study. All patients who were asked accepted and consented to be included in the investigation.

At the investigators hospital, insertion of pertitnoean dialysis catheters is performed by open surgery. This is performed using a three layer suture technique performed in local anesthesia. The technique enables immediate start of dialysis after surgery.

Outflow problems were defined as a delay of flow of more than 40 minutes for 500ml of PD fluid.

The duration of time was calculated by months on PD. Patients who died, were transplanted or changed for hemodialysis were censored. End-point was an insufficient drainage/flow of dialysis fluid that unabled adequate dialysis and intervention (by surgery) was necessary to correct/change catheter.

Statistical analyses used were Breslow test and Kaplan Meier survival curve.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients that are eligible and planned to start peritoneal dialysis and thereafter accept to be part of the study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-11; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
insufficient drainage/flow of dialysis fluid that unabled adequate dialysis | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ragnberth Helleday, MD, Study Chair — Medicincenter, Norrlands Universitetssjukhus, Umea, Sweden
Locations (1):
- Medicincenter, Norrlands Universitetssjukhus, Umeå, Sweden

REFERENCES:
- [Background] Di Paolo N, Capotondo L, Sansoni E, Romolini V, Simola M, Gaggiotti E, Bercia R, Buoncristiani U, Canto P, Concetti M, De Vecchi A, Fatuzzo P, Giannattasio M, La Rosa R, Lopez T, Lo Piccolo G, Melandri M, Vezzoli G, Orazi E, Pacitti A, Ramello A, Russo F, Napoli M, Tessarin MC. The self-locating catheter: clinical experience and follow-up. Perit Dial Int. 2004 Jul-Aug;24(4):359-64. PMID 15335150
- [Derived] Briggs VR, Jacques RM, Fotheringham J, Maheswaran R, Campbell M, Wilkie ME. Catheter insertion techniques for improving catheter function and clinical outcomes in peritoneal dialysis patients. Cochrane Database Syst Rev. 2023 Feb 22;2(2):CD012478. doi: 10.1002/14651858.CD012478.pub2. PMID 36810986
- [Derived] Stegmayr BG, Sperker W, Nilsson CH, Degerman C, Persson SE, Stenbaek J, Arnerlov C. Few Outflow Problems With a Self-locating Catheter for Peritoneal Dialysis: A Randomized Trial. Medicine (Baltimore). 2015 Dec;94(48):e2083. doi: 10.1097/MD.0000000000002083. PMID 26632891